CLINICAL TRIAL: NCT01603797
Title: Guided Internet-delivered Acceptance and Commitment Therapy for Chronic Pain Patients: a Randomized Controlled Trial
Brief Title: Guided Internet-delivered Acceptance and Commitment Therapy for Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerhard Andersson (Other Government)
Responsible Party: Sponsor-Investigator, Gerhard Andersson, Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: smartaSIAMB_GA
Record Dates: First submitted 2012-05-19; First posted 2012-05-22 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Pain
Keywords: internetdelivered CBT; chronic pain; acceptance and commitment therapy; mindfulness; guided self help
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet delivered ACT (Experimental): Internet delivered acceptance and commitment therapy (ACT), 7 weeks treatment
  Interventions: Behavioral: Guided internet-delivered acceptance and commitment therapy
- Online discussion forum (Active Comparator): Active wait-list condition. Were offered to participate in a moderated online discussion forum. After post-treatment assessment the control group were offered treatment.
  Interventions: Behavioral: Guided internet-delivered acceptance and commitment therapy

INTERVENTIONS:
Behavioral: Guided internet-delivered acceptance and commitment therapy — The treatment program consisted of seven sections and was based on ACT.The first part was about creative hopelessness and was followed in the next section by an introduction to willingness and to the process of acceptance of pain. Information and assignments about committed action and values were also part of the treatment program. Mindfulness exercises were a regular feature in the program. The last part was about how to maintain learned strategies but also an evaluation of the program.

SUMMARY:
The aim of this study was to investigate if guided internet-delivered acceptance and commitment therapy (ACT)would help chronic pain patients.

DETAILED DESCRIPTION:
The present study investigates internet-delivered ACT for persons with chronic pain. The use of internet as a delivery format for interventions could be a way of overcome many barriers (financial obstacles, reluctance to seek treatment and paucity of clinicians trained in ACT) that hinder persons with chronic pain to seek or receive adequate help. Persons were randomized to either treatment for 7 weeks or to a control group who were invited to participate in a moderated online discussion forum. Follow up data was collected six months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* that participants had undergone medical investigation (within one year)
* had regular access to the internet
* had functional impairment caused by chronic pain
* had internet access

Exclusion Criteria:

* ongoing medical investigations or treatment that could interfere with participation in the study, such as planned surgery and suffering from acute physical or psychological conditions
* not fluent in the Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Chronic Pain Acceptance Questionnaire (CPAQ) | One week pre- and post-treatment
  CPAQ consists of 20 items divided into two subscales: activity engagement and pain willingness. Items are rated on a scale from 0 (never true) to 6 (always true). Higher scores denote greater activity engagement and pain willingness. Studies show acceptable reliability (α =.72-.92).

SECONDARY OUTCOMES:
Hospital and Anxiety Depression Scale (HADS) | One week pre- and post- treatment
  HADS contains 14 items and evaluates severity of symptoms of depression and anxiety without contamination of scores of physical symptomatology.
The Coping Strategies Questionnaire (CSQ) | One week pre- and post- treatment
  The CSQ contains 50 items divided into eight scales measuring different cognitive and behavioural coping strategies and has been widely used by chronic pain patients. The coping strategies scales are: diverting attention, re-interpreting pain sensations, coping self-statements, ignoring sensations, praying and hoping, catastrophizing and increased behavioral activities
Multidimensional Pain Inventory (MPI-S) | One week pre- and post- treatment
  The Swedish version of MPI (MPI-S) consists of 34 items divided into 8 scales. The first section addresses: Pain Severity, Interference, Life Control, Affective Distress and Support. The second section addresses the patient's perception of how significant others respond to their displays of pain: Punishing Responses, Solicitous Responses and Distracting Responses.
The Pain and Impairment Relationship Scale (PAIRS) | One week pre- and post- treatment
  PAIRS assess beliefs and attitudes associated with the experience of chronic pain and one's ability to function despite pain. It consists of 15 personal statements that reflect thoughts, attitudes and opinions about pain.
Quality of Life Inventory (QOLI) | One week pre- and post- treatment
  QOLI consists of 32 items for assessing life satisfaction. The assessment yields an overall score and profile in 16 areas of life; health, self-esteem, goals and values, money, work, play, learning, creativity, helping, love, friends, children, relatives, home, neighborhood, and community.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Professor, Study Director — Linkoeping University; Monica Buhrman, MSc, Principal Investigator — Uppsala University; Timo Hursti, PhD, Study Chair — Uppsala University; Torsten Gordh, Professor, Study Chair — Uppsala University; Tomas Furmark, Professor, Study Chair — Uppsala University; Astrid Skoglund, MSc, Study Chair — Uppsala University; Josefin Husell, MSc, Study Chair — Uppsala University; Kristina Bergström, MSc, Study Chair — Uppsala University; Nina Bendelin, MSc, Study Chair — Linkoeping University

REFERENCES:
- [Derived] Bendelin N, Bjorkdahl P, Risell M, Nelson KZ, Gerdle B, Andersson G, Buhrman M. Patients' experiences of internet-based Acceptance and commitment therapy for chronic pain: a qualitative study. BMC Musculoskelet Disord. 2020 Apr 6;21(1):212. doi: 10.1186/s12891-020-03198-1. PMID 32252707